CLINICAL TRIAL: NCT03374592
Title: A Phase II Randomized Controlled Trial of Volumetric Intensity Modulated Arc Therapy vs. Conventional Radiotherapy for Cancer Pain
Brief Title: Volumetric Intensity Modulated Arc Therapy vs. Conventional Radiotherapy for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE14.046
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Neoplasm Metastasis; Pain; Radiotherapy Side Effect; Quality of Life
Keywords: Intensity-modulated radiation therapy; Volumetric intensity-modulated arc therapy; Radiotherapy; Pain; Metastasis; Quality of Life; Acute Toxicity
MeSH Terms: conditions — Neoplasm Metastasis; Pain; Radiation Injuries | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Radiotherapy (Active Comparator): 8Gy in 1 fraction or 20Gy in 5 fractions
  Interventions: Radiation: Conventional Radiotherapy
- Volumetric Intensity-Modulated Arc Therapy (Experimental): 8Gy in 1 fraction or 20Gy in 5 fractions
  Interventions: Radiation: Volumetric Intensity-Modulated Arc Therapy

INTERVENTIONS:
Radiation: Volumetric Intensity-Modulated Arc Therapy — Advanced radiotherapy technique
  Other Names: Intensity modulated radiotherapy
  Arms: Volumetric Intensity-Modulated Arc Therapy
Radiation: Conventional Radiotherapy — Conventional radiotherapy technique
  Arms: Conventional Radiotherapy

SUMMARY:
This study compares the use of conventional radiotherapy technique with volumetric intensity-modulated radiotherapy (VMAT) in the treatment of painful cancer metastases. Half of the patients will receive radiotherapy using a conventional technique, while the other half will receive their treatment using a the VMAT technique.

DETAILED DESCRIPTION:
Radiotherapy to painful sites of metastasis can provide pain relief.

Side-effects from radiotherapy is dependent on the volume and dose received by normal tissues. Conventional radiotherapy techniques delivers similar doses of radiation to the targeted cancer lesion and the normal tissues along the entrance and exit paths of the radiation.

Volumetric intensity-modulated arc therapy (VMAT) is an advanced technique of radiotherapy that spares normal tissues from receiving high-dose irradiation. However, VMAT increases the volume of normal tissues receiving low-dose irradiation.

This study aims at comparing the quality of life and side-effect profiles of patients treated by palliative radiotherapy using the conventional technique vs. VMAT.

ELIGIBILITY:
Inclusion Criteria:

1. Pain (SF-BPI score ≥1) should be related to metastases (bone or others) or to the tumor itself
2. Capable of providing the full list of analgesic medication being used
3. Capable of completing the SF-BPI and EORTC questionnaires without any help
4. Life expectancy of at least 3 month
5. KPS greater or equal to 50
6. Radiotherapy to 1 site pain
7. Site of treatment not previously irradiated
8. No planned changes in analgesic within 7 days before and after treatment

   • Patient may be started on Dexamethasone on the first day of radiotherapy
9. No planned chemotherapy, radiotherapy or surgery within 7 days before and after treatment
10. Patient provided informed consent to participate in this study

Exclusion Criteria:

1. Major mental or psychiatric impairments, which in the investigator's opinion will prevent administration or completion of the protocol therapy and/or interfere with follow-up.
2. Treatment to upper and lower limb
3. Treatment to 2 or more sites of pain
4. Re-irradiation of the site of treatment
5. Women who are pregnant
6. Life expectancy less than 3 month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QOL) | 1 week
  The global QOL subscale will be measured using the European Organization for Research and Treatment of Cancer (EORTC) QLQ C30 questionnaire and compared to baseline. The global QOL subscales will be scored according to the EORTC scoring manual (min: 0, max: 100). Higher scores represent better global QOL.

SECONDARY OUTCOMES:
Quality of Life - Function subscales | 3 month
  Quality of life function subscales (physical, role, cognitive, emotional, social and financial functions) will be measured using the European Organization for Research and Treatment of Cancer (EORTC) QLQ C30 questionnaire and compared to baseline. QOL subscales will be scored according to the EORTC scoring manual (min: 0, max: 100). For function subscales, higher scores represent better function.
Quality of Life - Symptom subscales | 3 month
  Quality of life symptom subscales (dyspnea, pain, fatigue, appetite loss, nausea, constipation, and diarrhea symptoms) will be measured using the European Organization for Research and Treatment of Cancer (EORTC) QLQ C30 questionnaire and compared to baseline. QOL subscales will be scored according to the EORTC scoring manual (min: 0, max: 100). For symptom subscales, higher scores represent worse symptoms.
Pain relief | 1 week
  Pain response to radiotherapy as defined by the International Bone Metastases Consensus Endpoint Definitions
Pain relief | 1 month
  Pain response to radiotherapy as defined by the International Bone Metastases Consensus Endpoint Definitions
Pain relief | 3 month
  Pain response to radiotherapy as defined by the International Bone Metastases Consensus Endpoint Definitions
Toxicities | 1 week
  Descriptive tabulation of toxicities related to radiotherapy as defined by CTCAE v4
Toxicities | 1 month
  Descriptive tabulation of toxicities related to radiotherapy as defined by CTCAE v4
Toxicities | 3 month
  Descriptive tabulation of toxicities related to radiotherapy as defined by CTCAE v4

OTHER OUTCOMES:
Resource utilization | Baseline
  Time spent in planning and delivering radiotherapy
Physical activity | 1 week
  Change in the daily number of steps taken by patients before and after radiotherapy as measured using an activity tracker
Blood biomarkers | 1 week
  Change in cytokine levels in blood following radiotherapy as a biomarker of response to radiotherapy
Blood biomarkers | 1 week
  Change in circulating microRNA levels in blood following radiotherapy as a biomarker of response to radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wong, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wong P, Lambert L, Thanomsack P, Coulombe G, Lambert C, Charpentier AM, Barkati M, Fortin I, Lafontaine J, Roberge D. Quality of Life: A Prospective Randomized Trial of Palliative Volumetric Arc Therapy Versus 3-Dimensional Conventional Radiation Therapy. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1431-1439. doi: 10.1016/j.ijrobp.2020.11.061. Epub 2020 Nov 28. PMID 33259935
- [Result] Dorion V, Lambert L, Frazzi A, Cayer JF, Wong P. A Pilot Study in the Use of Activity Trackers for Assessing Response to Palliative Radiotherapy. Cureus. 2017 Nov 22;9(11):e1871. doi: 10.7759/cureus.1871. PMID 29383293